CLINICAL TRIAL: NCT03592563
Title: CUHK Brain Health Longitudinal Study
Acronym: BHS
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Leung Wai Hong Thomas, Professor, Chinese University of Hong Kong
Other Study IDs: Crec No. 2018.148
Record Dates: First submitted 2018-06-13; First posted 2018-07-19 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Stroke, Ischemic; Stroke Syndrome; Stroke; Stroke, Acute; Dementia; Brain Ischemia; Brain Diseases; Alzheimer Disease; Health Attitude; Health Knowledge, Attitudes, Practice; Health Personnel Attitude; Healthy Aging
Keywords: stroke; dementia; Alzheimer disease; Health Brain; Health knowledge
MeSH Terms: conditions — Ischemic Stroke; Stroke; Dementia; Brain Ischemia; Brain Diseases; Alzheimer Disease; Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 30ml of EDTA blood will be collected for genome sequencing or PCR gene expression.
  5-10ml of stool will be collected for microbiome study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Red group: Those participants who had established diagnosis of one or more neurological and/or psychiatric conditions
  Baseline: The participants' medical history, signs, symptoms and diagnoses of neurological and/or psychiatric disorders would be recorded. Neuro-QoL questionnaire plus an additional subset of questions based on their clinical diagnosis should be done.
  Interventions: Behavioral: Neuro-QoL questionnaire
- Yellow group: Those participants who are high-risk to develop one or more neurological and/or psychiatric conditions, for example:
  1. family history (first degree relative) one or more neurological and/or psychiatric conditions;
  2. examination, imaging or laboratory findings consistent with pre-symptomatic stages of one or more neurological and/or psychiatric disorders.
  Baseline: The participants' medical history, signs, symptoms and diagnoses of neurological and/or psychiatric disorders would be recorded. Neuro-QoL questionnaire should be done.
  Interventions: Behavioral: Neuro-QoL questionnaire
- Green group: Those participants who are not meeting criteria for Red or Yellow groups, but interested in longitudinal research on maintenance and/or improvement of their brain health.
  Baseline: The participants' medical history would be recorded and Neuro-QoL questionnaire should be done.
  Interventions: Behavioral: Neuro-QoL questionnaire

INTERVENTIONS:
Behavioral: Neuro-QoL questionnaire — Follow-up over time will continue (either in-person or over the phone) using the same questionnaires (depending on which group they are belongs to) at approximately 6-month intervals. During each follow-up, participants will be screened for any new signs, symptoms and diagnoses of neurological and/or psychiatric disorders, in order to correlate these outcomes with risk factors captured using the procedures described above.

SUMMARY:
The goal of this study is to develop a large longitudinal cohort of individuals diagnosed with or at high risk for brain diseases (both neurological and psychiatric in nature), in order to identify risk factors that contribute to neurological and psychiatric diseases over time. The investigators seek to capture relevant information from medical records, electronically administered questionnaires and follow up phone-based interviews. The investigators expect to eventually have sufficient power from our dataset to examine risk factors for a variety of brain disorders, both individually and in aggregate. Our ultimate goal is to offer scientifically validated ways to preserve and promote brain health by working with our patients' needs and tracking their progress over time.

DETAILED DESCRIPTION:
For those interested participants, our services coordinator, co-investigator or principal investigator will interview and explain the study in detail and obtain your consent. After signed the consent, the participant should complete the Neuro-QoL (Quality of Life in Neurological Disorders) questionnaire first, either on-site at CUHK Brain Health Centre located at Tsim Sha Tsui in Hong Kong, PWH or community centre. The questions in the questionnaire focus on the following: ability to participate in social roles, emotional and behavioral dyscontrol, fatigue, lower extremity function, stigma, upper extremity function, positive affect and well-being, satisfaction with social roles, cognitive function, anxiety and depression. These questions enable us to get a full picture of the participant's health. Participants in Green and yellow groups will receive this standard battery of questions. However, participants in Red group may receive an additional subset of questions based on their clinical diagnosis. Once again, all subjects are asked to complete this questionnaire for clinical evaluation purposes, regardless of whether or not they decide to participate in this study.

When the participant is willing to join the study, an evaluation would be scheduled. At that visit, our physician and/or study coordinator will review the participant's medical history, current concerns, and responses to the questionnaires. Diagnostic and therapeutic recommendations may be offered, as warranted. The investigator or physician will determine whether a follow-up clinic visit is warranted. Depending on the physician's recommendations, the participant will either participate in a research phone call in approximately 6 months, or will be scheduled for in person research follow up. In addition to the phone call or clinic visit, and will also receive an identical questionnaire to the first one by e-mail, by phone, or in person. Follow-up over time will continue (either in-person or over the phone) using the same questionnaires at approximately 6-month intervals. During follow-up, participant will be screened for new signs, symptoms and diagnoses of neurological and/or psychiatric disorders, in order to correlate these outcomes with risk factors captured using the procedures described above.

The proposed study does not involve formulating new diagnoses or directly offering treatment for neurological and/or psychiatric conditions. All patients admitted to PWH or other medical institutes will be treated according to the standard care at the corresponding institution, regardless of their decision to participate in this repository. Should results from this study lead to discovery of one or more factors associated with development of brain disease, the principal investigators, co-investigators, or study coordinator in the CUHK Brain Health Centre will inform, counsel and offer diagnostic and/or therapeutic recommendations to participants accordingly. The participants may be referred to relevant departments for follow-up clinical visits and may also be invited to participate in sister research projects at PWH/CUHK that have obtained ethics approval; if the participants are interested in any sister projects, they may be offered tests as the study procedures of these projects, including but not limited to blood tests, genetic tests, retinal imaging and brain imaging exams.

Our study aims to follow longitudinally individuals with or at risk for neurological and psychiatric disease, regardless of gender or sexual orientation. The investigators focus on enrolling adults as the vast majority of the neurological and psychiatric conditions of interest are diagnosed well into adulthood; indeed, most are age-related and particularly frequent among individuals in the fifth decade of life and beyond. Our study uniquely welcomes even individuals who are healthy from a brain standpoint, and offers them an opportunity to increase our scientific understanding of the early transition from normal to pathological brain functioning. As a result, the entire population as a whole stand to potentially benefit from the outcomes of the proposed research.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years of age
2. Fulfilling criteria for membership in one of these three groups:

   * Red group: established diagnosis of one or more neurological and/or psychiatric conditions
   * Yellow group: high-risk to develop one or more neurological and/or psychiatric conditions

     1. family history (first degree relative) one or more neurological and/or psychiatric conditions
     2. examination, imaging or laboratory findings consistent with pre-symptomatic stages of one or more neurological and/or psychiatric disorders
   * Green group: not meeting criteria for Red or Yellow groups, but interested in longitudinal research on maintenance and/or improvement of brain health
3. Subject provides informed consent by signing and dating the written informed consent form
4. Subject is willing to answer health questionnaires and be followed longitudinally

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Chinese ONLY
  2. Hong Kong Resident
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2038-12-31 (Estimated); Study Completion 2048-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk factors contributing to neurological and psychiatric diseases | December, 2038
  The participants' electronic medical records and questionnaires done (either symptomatic or asymptomatic) would be compared with their follow-up electronic medical records/phone follow-up interview and questionnaires done over time.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wai Hong LEUNG, FRCP, Principal Investigator — Division of Neurology, The Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Chinese University of Hong Kong, Hong Kong
  - The Chinese University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and health information may be sent out to our research collaborators at Massachusetts General Hospital and Harvard Medical School, where there is a sister institute for brain health for additional analysis.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The de-identified health information and data would be stored for more than 10 years, so that we can offer scientifically validated ways to preserve and promote brain health by working with our patients' needs and tracking their progress over time. This is because individuals diagnosed with neurological and psychiatric disorders can experience the very first symptoms up to 10-20 years before diagnosis.
Access Criteria: These de-identified data will be stored by collaborating institutions in a manner consistent with data storing secure procedures. Only principle investigator, study coordinator and related staffs can access.